CLINICAL TRIAL: NCT06596265
Title: Community Park-Based Programs for Health Promotion: The Fit2Lead Prospective Cohort Study
Acronym: F2L
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Miami-Dade County Parks and Recreation (Other); The Children's Trust, Miami FL (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105669_2
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Wellness, Psychological; Overweight or Obesity; Hypertension; Prehypertension; Low Physical Fitness
Keywords: Youth; Adolescent; Afterschool; Parks and Recreation; Mental Health; Physical Helath; Resilience; Violence Prevention
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being; Overweight; Obesity; Hypertension; Prehypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fit2 Lead Cohort 1-2: Fit2Lead runs September through June at no charge, and provides daily academic support, sports and recreation, meditation, stress resilience, and life skills-focused workshops. Participants who reach age 15 years and are awaiting an internship placement can remain in phase 1 until a position opens or can be transferred to another internship program within the MDPROS.
  Interventions: Behavioral: Fit2Lead Group 1-2

INTERVENTIONS:
Behavioral: Fit2Lead Group 1-2 — Each park serves anywhere from 2 to 9 feeder schools within these neighborhoods (a target population of 34 000 youth residents aged 12-17 years), and transportation from schools to parks is provided at no cost within a 3-mile radius of a program park. Fit2Lead participants can also enroll in the MDPROS youth summer camp at no charge.
  Work assignments support MDPROS operations and recreation staff. Interns in Phase II rotate every 8 weeks for exposure to different job opportunities, supervisors, and mentors.
  Duke is conducting a secondary data analysis on data collected as part of the Fit2Lead study.

SUMMARY:
The Fit2Lead prospective cohort study examines the effects of a park-based youth mental health and resilience afterschool program on youth participant mental health, resilience, physical fitness, and violence prevention outcomes. Duke will perform a secondary analysis of the data collected as part of the Fit2Lead prospective cohort study run by Miami-Dade County Parks and Recreation.

DETAILED DESCRIPTION:
The Fit2Lead prospective cohort study examines the effects of a park-based youth mental health and resilience afterschool program on youth physical and mental health and resilience, communication, and problem-solving skills training for underserved youth aged 12 to 17 years through an interdisciplinary collaboration among Miami-Dade Department of Parks, Recreation and Open Spaces (MDPROS) Miami-Dade County (MDC) Juvenile Services Department, MDC Public Schools, MDC Police Department, University of Miami, Florida International University, and other community-based partners.

Fit2Lead consists of 2 phases initiated simultaneously in 2015. For youth aged 12 to 14 years, Fit2Lead is offered after school Monday through Friday from 3:00 pm to 7:00 pm at 12 MDC parks for participants in under resourced neighborhoods and based on area-level youth crime and neighborhood poverty. Fit2Lead runs September through June at no charge, and provides daily academic support, sports and recreation, meditation, stress resilience, and life skills-focused workshops. Each park serves anywhere from 2 to 9 feeder schools within these neighborhoods (a target population of 34 000 youth residents aged 12-17 years), and transportation from schools to parks is provided at no cost within a 3-mile radius of a program park. Fit2Lead participants can also enroll in the MDPROS youth summer camp at no charge.

Phase II of Fit2Lead is for youth aged 15 to 17 years and entails a year-round paid internship and 3-hour weekly enrichment, resilience, and life skills workshops. Daily entry-level part-time interns receive $9 per hour (approximately 500 total paid hours per year; total salary approximately $4000 per participant, per year). Work assignments support MDPROS operations and recreation staff. Interns rotate every 8 weeks for exposure to different job opportunities, supervisors, and mentors. Phase 1 participants who reach age 15 years and are awaiting an internship placement can remain in phase 1 until a position opens or can be transferred to another internship program within the MDPROS.

ELIGIBILITY:
Inclusion Criteria:

* All participants enrolled in the Miami-Dade Fit2Lead study will be included in this secondary analysis
* Aged 12-17 years, residing in Miami-Dade County

Exclusion Criteria:

* Anyone not enrolled in the Miami-Dade Fit2Lead study will be excluded from this secondary analysis
* Aged <12 or >17 years, not residing in Miami-Dade County, cannot read and speak in English

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fit2Lead is offered in areas composed of 48% male youths, 60% Hispanic persons, 29% non-Hispanic Black persons, 33% single-parent households, and 33% of residents living below the federal poverty threshold as defined by the American Community Survey. Thirty-three percent of families are single-parent households, and 33% of residents are living in poverty in zip codes where Fit2Lead is offered.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-02-17 (Actual); Primary Completion 2028-06-17 (Estimated); Study Completion 2028-06-17 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | Baseline, 12-72 months
Change in Blood Pressure | Baseline, 12-72 months
Change in number of push-ups | Baseline, 12-72 months
Change in number of sit-ups | Baseline, 12-72 months
Change in Career and Education Planning survey | Baseline, 12-72 months
Change in College and Career Readiness survey | Baseline, 12-72 months
Change in Kidscreen-27 | Baseline, 12-72 months
  The Kidscreen-27 score range is 27-135. A higher score indicates more positive well-being.
Change in Generalized Anxiety Disorder 7-item (GAD-7) | Baseline, 12-72 months
  The GAD-7 has a score range 0-21. Higher score indicates higher anxiety levels.
Change in Patient Health Questionnaire-8 (PHQ-8) | Baseline, 12-72 months
  The PHQ-8 has a score range 0-24. Higher score indicates higher depression levels.
Change in the Progressive Aerobic Cardiovascular Endurance Run (PACER) score | Baseline, 12-72 months
  Among boys, for ages 10-17, the healthy fitness range is 23-61 laps for age 10, 23-72 laps for age 11, 32-72 laps for age 12, and 41-83 laps for ages 13 and up; Among girls, for ages 10-17, the healthy fitness range is 7-41 laps for age 10, 15-41 laps for ages 11 and 12, and 23-51 laps for ages 13 and up. A higher score indicates greater aerobic capacity.
Change in Brief Sense of Community Scale (BSCS) | Baseline, 12-72 months
  The Brief Sense of Community Scale (BSCS) has a total score range of 0-32. Higher score indicates more positive sense of community.
Change in Sociopolitical Control Scale for Youth (SCPS-Y; Leadership subscale) | Baseline, 12-72 months
  The SCPS-Y has a range 1-6. Higher scores indicate higher policy control, leadership competence, sense of community, ethnic identity, and social support.
Change in Self-efficacy for teen conflict (SE-TCS) | Baseline, 12-72 months
  Possible range for the SE-TCS is 5 to 25' with higher scores indicating more confidence
Change in Casey Life Skills Assessment | Baseline, 12-72 months
  Casey Life Skills Assessment (CLSA) scores are on a scale of 1-5, with 5 representing the highest level of strength
Change in Perceived Stress Scale (PSS) | Baseline, 12-72 months
  The Perceived Stress Scale (PSS) has a score range of 0 to 40, with higher scores indicating greater perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Emily D'Agostino, Principal Investigator — Duke University
Locations (1):
- Miami-Dade County Parks, Recreation and Open Spaces Department, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Agostino EM, Frazier SL, Hansen E, Patel HH, Ahmed Z, Okeke D, Nardi MI, Messiah SE. Two-Year Changes in Neighborhood Juvenile Arrests After Implementation of a Park-Based Afterschool Mental Health Promotion Program in Miami-Dade County, Florida, 2015-2017. Am J Public Health. 2019 Jun;109(S3):S214-S220. doi: 10.2105/AJPH.2019.305050. PMID 31241997
- [Background] D'Agostino E, Frazier SL, Hansen E, Nardi MI, Messiah SE. Association of a Park-Based Violence Prevention and Mental Health Promotion After-School Program With Youth Arrest Rates. JAMA Netw Open. 2020 Jan 3;3(1):e1919996. doi: 10.1001/jamanetworkopen.2019.19996. PMID 31995210
- [Background] Goodman AC, Ouellette RR, D'Agostino EM, Hansen E, Lee T, Frazier SL. Promoting healthy trajectories for urban middle school youth through county-funded, parks-based after-school programming. J Community Psychol. 2021 Sep;49(7):2795-2817. doi: 10.1002/jcop.22587. Epub 2021 Apr 29. PMID 33914915
- [Background] Frazier SL, Chou T, Ouellette RR, Helseth SA, Kashem ER, Cromer KD. Workforce Support for Urban After-School Programs: Turning Obstacles into Opportunities. Am J Community Psychol. 2019 Jun;63(3-4):430-443. doi: 10.1002/ajcp.12328. Epub 2019 Apr 19. PMID 31002394
- [Background] Cromer KD, D'Agostino EM, Hansen E, Alfonso C, Frazier SL. After-school poly-strengths programming for urban teens at high risk for violence exposure. Transl Behav Med. 2019 May 16;9(3):541-548. doi: 10.1093/tbm/ibz013. PMID 31094433